CLINICAL TRIAL: NCT05041283
Title: Impact of Artificial Intelligence-based Patient Reinforcement on Quality of Colonoscopy
Acronym: ARCHES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Prof. Dr. med., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ARCHES
Record Dates: First submitted 2021-09-06; First posted 2021-09-13 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Bowel Preparation
Keywords: Bowel Preparation; Artificial Intelligence; Polyp Detection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Preparation (No Intervention): Control arm; patients receive a standard support for bowel preparation consisting of a explanatory dialogue with a gastroenterologist and a brochure with a structurated description of bowel preparation and colonoscopy conduct
- Phone-call Supported Preparation (Active Comparator): In addition to standard preparation, patients receive a phone call every day starting at 3 days before colonoscopy in which a investigator explains key points of bowel preparation and patients can ask questions concerning bowel preparation and colonoscopy conduct.
  Interventions: Other: Phone call
- Chatbot Supported Preparation (Experimental): In addition to standard preparation, patients receive an access to a chatbot which can be contacted via Whats App starting at 3 days before colonoscopy. The chatbot is programed to answer questions concerning bowel preparation and colonoscopy conduct.
  Interventions: Other: Chatbot

INTERVENTIONS:
Other: Chatbot — A artificial-intelligence based chatbot is provided 3 days before colonoscopy to answer questions concerning bowel preparation and colonoscopy conduct.
  Arms: Chatbot Supported Preparation
Other: Phone call — A phone call is performed every day starting at 3 days before colonoscopy to support bowel preparation.
  Arms: Phone-call Supported Preparation

SUMMARY:
In order to improve bowel preparation for colonoscopy and consequently enhance detection rate of malignant and premalignant findings, a prospective, randomized and controlled three-arm study was developed. Patients who undergo ambulatory colonoscopy are randomly assigned into a control group with standard preparation, a phone call supported preparation group or a group supported by an artificial intelligence based chatbot. Primary endpoint is defined as quality of bowel preparation (Boston Bowel Preparation Score), secondary endpoints are patients satisfaction, comprehensiveness of bowel preparation, sedation dose, rate of coecal intubation and the rate of adenoma and polyp detection, anxiety referred to colonoscopy and patients satisfaction with preparation support.

DETAILED DESCRIPTION:
Adequate bowel preparation is crucial for detection of adenoma and polyps of the colon, which can transform into malignant and premalignant lesions. In particular ambulatory performed colonoscopy is often insufficient due to inadequate preparation by patients at home. To focus this issue, a artificial intelligence based chatbot was developed to help patients who undergo bowel preparation by answering questions concerning bowel preparation. To compare the effect of this program, a three-arm randomized, controled multicentric clinical trial was developed. All patients who undergo ambulatory colonoscopy and meet the inclusion criteria (18 y.o., informed consent, WhatsApp access) were randomized in a standard preparation group (medical briefing and preparation brochure), a group receiving phone calls with instructions for bowel preparation and a third group with access to the chat bot answering questions concerning bowel preparation and examination conduct. As the primary end point, the quality of bowel preparation measured as Boston Bowel Preparation Scale was defined. As secondary endpoints patients satisfaction, comprehensiveness of bowel preparation, sedation dose, rate of coecal intubation, the rate of adenoma and polyp detection, anxiety referred to colonoscopy and patients satisfaction with preparation support were measured.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* smartphone with access to WhatsApp
* indication for ambulatory colonoscopy
* ASA I or II

Exclusion Criteria:

* no informed consent given or possible
* no access to a smartphone with WhatsApp
* <18 years old
* Pregnancy/Lactation
* Allergy to Moviprep©
* ASA (American Society of Anesthesiologists) state >II
* extended abdominal surgery in past history
* no indication for ambulatory colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel preparation | During colonoscopy
  evaluated with the Boston Bowel Preparation Scale (0-9, 1=worst preparation, 9= best preparation)

SECONDARY OUTCOMES:
Patients satisfaction with bowel preparation | Immediately after the intervention
  Via questionnaire; 8 items, ordinal scale with 4 grades (completely satisfied/mainly satisfied/mainly dissatisfied/completely dissatisfied)
Comprehensiveness of bowel preparation | During colonoscopy
  Rate of successfully completed colonoscopy without premature termination due to remaining feces(from anus to terminal ileum)
Sedation dose | During colonoscopy
  Total amount of administered sedation per examination
Coecal intubation | During colonoscopy
  Successful coecal intubation during colonoscopy
Polyp and adenoma detection rate | During colonoscopy
  Rate of detected polyps and adenomas
Patients satisfaction with preparation support | Within 3 days after the intervention
  Via questionnaire; 8 items, ordinal scale with 4 grades (completely satisfied/mainly satisfied/mainly dissatisfied/completely dissatisfied)
Anxiety referred to colonoscopy | Within 3 days before the intervention and 3 days after the intervention; 8 items with binary answer yes/no)
  German ABI-MS questionnaire (questionnaire on overcoming fear considering medical therapy;

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, Prof., Principal Investigator — University Hospital Ulm
Locations (3):
- Germany (3):
  - Specialist Practice Profes. Dikopoulos/Ludwig, Ulm, Baden-Würrtemberg
  - University of Ulm, Interdisciplinary Endoscopy, Ulm, Baden-Würrtemberg
  - Specialist Practice, Berlin